CLINICAL TRIAL: NCT05009849
Title: Randomized Controlled Evaluating the Role of Exercise in Women Undergoing Treatment for Breast Cancer
Brief Title: Role of Exercise in Breast Cancer Patient Undergoing Treatment
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tata Memorial Centre (Other)
Responsible Party: Principal Investigator, Nita Sukumar Nair, Professor and Surgeon (Breast Surgical Oncology Services), Tata Memorial Centre
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 735
Record Dates: First submitted 2021-07-29; First posted 2021-08-18 (Actual); Last update posted 2022-10-20 (Actual); Status verified 2022-10

CONDITIONS: Breast Cancer Patients

STUDY DESIGN:
Intervention Model Description: Arm I: Yoga & Conventional Exercises Arm II: Conventional Exercises All eligible patients will be randomly to either of the arm as mentioned above.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise I (Experimental): Yogic and Routine Exercises (referred to as exercise I) Phase I: 1-7 days (Minimum attendance 4 days), Phase II: 8 - 14 days (Minimum attendance 4 days), Phase III: at 6-9 months or 12-15 months 1 year up gradation of exercises at 6-9 month or 12-15 months 1 year (Depending upon compliance to phase II exercises) Objective assessment at baseline, 14 days, 6-9, 12-15, 18-21, 36-39 and 54-57 months Exercise evaluation will be done at 6-9, 12-15, 30-33, 48-51 and 66-69 months
  Interventions: Other: Yoga Exercises
- Exercise II (Active Comparator): Objective assessment at baseline, 14 days, 6-9, 12-15, 18-21, 36-39 and 54-57 months
  Interventions: Other: Yoga Exercises

INTERVENTIONS:
Other: Yoga Exercises — The exercises in the Exercise I arm (Yoga and conventional exercises) will be upgraded to Phase II. Patients will be allowed to attend a minimum of four out of seven days in Phase I and II. Patients will be assessed at 6-9 months for compliance to phase II exercises. Only if patients are fulfilling the criteria for accuracy, sequence and duration of phase II exercises, will they be taught phase III exercises. Patients who are unable to do phase II exercises accurately or demonstrate non compliance to the exercise routine at first follow up visit/ 6-9 months will be re taught phase II exercises. These patients will be upgraded to phase III only if able to perform phase II adequately at assessment. Six months after completion of phase III exercises, patients will be assessed for compliance to phase III exercises. These women's will be assessed at the subsequent 6-9 month follow up and compliance will be evaluated.

SUMMARY:
Randomized controlled trial to evaluate the impact of yoga on QOL is also powered to evaluate the impact of yoga on survival. Study involves various phases of yoga(divided in three phases: Phase I/II/III) during treatment and survivorship, with a comparative analysis of different time points and the response to yoga, which will help integrating yoga as a complementary modality. Also, this study will help identify the long term and short term effects of this therapy in breast cancer patients and survivors.

One of the main differences between yoga and other forms of physical activity is that yoga exercises oppose violent muscle movement and is designed to counteract fatigue through relaxation and breathing. 6 monthly Follow Up will be for 5 years followed by yearly follow up.

DETAILED DESCRIPTION:
Women with breast cancer are constantly exploring measures in addition to ongoing conventional therapy to relieve disease related symptoms, minimize side effects associated with conventional treatment, reduce their risk of recurrence and enhance their prospects for survival. Breast cancer survival rates have considerably improved over the years with the advent of new therapeutic measures and early detection. However its treatment sequelae are associated with significant changes in quality of life (QOL) and well being. Fatigue is one of the most prevalent QOL concerns, affecting 30% to 70% of breast cancer survivors.

Yoga is based on the practice of physical postures, breathing techniques and meditation. Philosophically, it aims at increasing the body's ability to master the mind with the goal of spiritual awareness and connection. A randomized trial of yoga in women with breast cancer undergoing radiation therapy demonstrated an improvement in impact of events scale at 3 months suggesting that the more intrusive thoughts at 1 month the greater the finding of meaning in cancer by 3 months.

* This is the first randomized controlled trial of this magnitude (850 women), which in addition to testing the impact of yoga on QOL is also powered to evaluate the impact of yoga on survival
* This is a longitudinal study measuring various phases of yoga during treatment and survivorship, with a comparative analysis of different time points and the response to yoga , which will help integrating yoga as a complementary modality
* Also, this study will help identify the long term and short term effects of this therapy in breast cancer patients and survivors
* The exercises are carefully designed keeping the phase of treatment or recovery of the breast cancer patient/survivor in focus.
* Chronic ailments have also been kept in mind (eg: which impede mobility or flexibility ie: spondylosis)
* One of the main differences between yoga and other forms of physical activity is that yoga exercises oppose violent muscle movement and is designed to counteract fatigue through relaxation and breathing.

ELIGIBILITY:
Inclusion Criteria:

* Women with unilateral breast cancer
* Age 18-65 years

Exclusion Criteria:

* Metastatic breast cancer
* Pregnant Women
* Women with physical limitations to perform exercises
* Previous history of cancer

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Womens with breast Cancer
Enrollment: 850 (Actual)
Dates: Start 2010-11-23 (Actual); Primary Completion 2025-05-24 (Estimated); Study Completion 2030-05-30 (Estimated)

PRIMARY OUTCOMES:
Disease-free survival | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 60 months.
  To assess the effect of yoga on disease free survival in women breast cancer.

SECONDARY OUTCOMES:
Assess the impact of Yoga on inflammatory cytokines and cell free chromatin | From randomization to 12 months
  The impact of yoga on inflammatory markers will be assessed by using serum samples to check the concentration of IL2, TNF alpha, IL6, IL8, IL10 and C reactive protein by using ELISA technique.
Pain assessment | from randomization to 60 months
  To assess the effect of yoga using Pain Assessment chart questionnaire, having score scale from scale 0 to 10 wherein 0 represent "No Pain" and 10 represent "Worst Possible Pain"
Quality of life assessment | from randomization to 60 months
  To assess the effect of yoga using Quality of life questionnaire (QLQ-30, BR-23, Spirituality & BFI having score scale from 1-4, wherein 1 represents 'Not at All' and 4 'very much'
Improvements in Lung Function | The FEV1/ FVC ratio and the value will be checked, if the value is within 80% to 120%, it will be considered as normal (95 percent confidence interval). From randomization until 12 months.
  To assess the effect of yoga in improving the Lung Function by evaluating Pulmonary Function Teast (PFT) readings.
Improvements in Overall survival | from the date of randomization to the date of death or censored at the date of last follow up for the patients who are alive or lost to follow up, until 60 months
  To assess the effect of yoga on overall free survival in women breast cancer.

CONTACTS AND LOCATIONS:
Overall Officials: nita nair, Mch, Principal Investigator — Tata Memorial Centre

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Knols R, Aaronson NK, Uebelhart D, Fransen J, Aufdemkampe G. Physical exercise in cancer patients during and after medical treatment: a systematic review of randomized and controlled clinical trials. J Clin Oncol. 2005 Jun 1;23(16):3830-42. doi: 10.1200/JCO.2005.02.148. PMID 15923576
- [Background] Lemieux J, Topp A, Chappell H, Ennis M, Goodwin PJ. Economic analysis of psychosocial group therapy in women with metastatic breast cancer. Breast Cancer Res Treat. 2006 Nov;100(2):183-90. doi: 10.1007/s10549-006-9249-1. Epub 2006 Jun 14. PMID 16773438
- [Background] Jones SB, Thomas GA, Hesselsweet SD, Alvarez-Reeves M, Yu H, Irwin ML. Effect of exercise on markers of inflammation in breast cancer survivors: the Yale exercise and survivorship study. Cancer Prev Res (Phila). 2013 Feb;6(2):109-18. doi: 10.1158/1940-6207.CAPR-12-0278. Epub 2012 Dec 4. PMID 23213072
- [Background] L. Cohen, K. D. Chandwani, G. Perkins, B. Thornton, B. Arun, N. V. Raghuram, H. R. Nagendra Randomized trial of yoga in women with breast cancer. Undergoing radiation treatment: Long-term effects. J Clin Oncol 26: 2008 (May 20 suppl; abstr 9639).
- [Result] Newman V, Rock CL, Faerber S, Flatt SW, Wright FA, Pierce JP. Dietary supplement use by women at risk for breast cancer recurrence. The Women's Healthy Eating and Living Study Group. J Am Diet Assoc. 1998 Mar;98(3):285-92. doi: 10.1016/s0002-8223(98)00068-6. PMID 9508010
- [Result] Risberg T, Lund E, Wist E, Kaasa S, Wilsgaard T. Cancer patients use of nonproven therapy: a 5-year follow-up study. J Clin Oncol. 1998 Jan;16(1):6-12. doi: 10.1200/JCO.1998.16.1.6. PMID 9440716
- [Result] Beisecker A, Cook MR, Ashworth J, Hayes J, Brecheisen M, Helmig L, Hyland S, Selenke D. Side effects of adjuvant chemotherapy: perceptions of node-negative breast cancer patients. Psychooncology. 1997 Jun;6(2):85-93. doi: 10.1002/(SICI)1099-1611(199706)6:23.0.CO;2-T. PMID 9205966
- [Result] Wallgren A. Late effects of radiotherapy in the treatment of breast cancer. Acta Oncol. 1992;31(2):237-42. doi: 10.3109/02841869209088909. PMID 1622640
- [Result] Gyenes G, Fornander T, Carlens P, Rutqvist LE. Morbidity of ischemic heart disease in early breast cancer 15-20 years after adjuvant radiotherapy. Int J Radiat Oncol Biol Phys. 1994 Mar 30;28(5):1235-41. doi: 10.1016/0360-3016(94)90500-2. PMID 8175411
- [Result] Irvine D, Brown B, Crooks D, Roberts J, Browne G. Psychosocial adjustment in women with breast cancer. Cancer. 1991 Feb 15;67(4):1097-117. doi: 10.1002/1097-0142(19910215)67:43.0.co;2-z. PMID 1991258
- [Result] Coleman MP, Rachet B, Woods LM, Mitry E, Riga M, Cooper N, Quinn MJ, Brenner H, Esteve J. Trends and socioeconomic inequalities in cancer survival in England and Wales up to 2001. Br J Cancer. 2004 Apr 5;90(7):1367-73. doi: 10.1038/sj.bjc.6601696. PMID 15054456
- [Result] Burgess C, Cornelius V, Love S, Graham J, Richards M, Ramirez A. Depression and anxiety in women with early breast cancer: five year observational cohort study. BMJ. 2005 Mar 26;330(7493):702. doi: 10.1136/bmj.38343.670868.D3. Epub 2005 Feb 4. PMID 15695497
- [Result] Kornblith AB, Ligibel J. Psychosocial and sexual functioning of survivors of breast cancer. Semin Oncol. 2003 Dec;30(6):799-813. doi: 10.1053/j.seminoncol.2003.08.025. PMID 14663780
- [Result] Shapiro SL, Lopez AM, Schwartz GE, Bootzin R, Figueredo AJ, Braden CJ, Kurker SF. Quality of life and breast cancer: relationship to psychosocial variables. J Clin Psychol. 2001 Apr;57(4):501-19. doi: 10.1002/jclp.1026. PMID 11255204
- [Result] Mols F, Vingerhoets AJ, Coebergh JW, van de Poll-Franse LV. Quality of life among long-term breast cancer survivors: a systematic review. Eur J Cancer. 2005 Nov;41(17):2613-9. doi: 10.1016/j.ejca.2005.05.017. Epub 2005 Oct 13. PMID 16226458
- [Result] Arndt V, Merx H, Sturmer T, Stegmaier C, Ziegler H, Brenner H. Age-specific detriments to quality of life among breast cancer patients one year after diagnosis. Eur J Cancer. 2004 Mar;40(5):673-80. doi: 10.1016/j.ejca.2003.12.007. PMID 15010067
- [Result] Cella D, Fallowfield L, Barker P, Cuzick J, Locker G, Howell A; ATAC Trialistsa9 Group. Quality of life of postmenopausal women in the ATAC ("Arimidex", tamoxifen, alone or in combination) trial after completion of 5 years' adjuvant treatment for early breast cancer. Breast Cancer Res Treat. 2006 Dec;100(3):273-84. doi: 10.1007/s10549-006-9260-6. Epub 2006 Jun 21. PMID 16944295
- [Result] Vacek PM, Winstead-Fry P, Secker-Walker RH, Hooper GJ, Plante DA. Factors influencing quality of life in breast cancer survivors. Qual Life Res. 2003 Aug;12(5):527-37. doi: 10.1023/a:1025098108717. PMID 13677497
- [Result] Ganz PA, Guadagnoli E, Landrum MB, Lash TL, Rakowski W, Silliman RA. Breast cancer in older women: quality of life and psychosocial adjustment in the 15 months after diagnosis. J Clin Oncol. 2003 Nov 1;21(21):4027-33. doi: 10.1200/JCO.2003.08.097. PMID 14581426
- [Result] Courneya KS, Friedenreich CM, Sela RA, Quinney HA, Rhodes RE, Handman M. The group psychotherapy and home-based physical exercise (group-hope) trial in cancer survivors: physical fitness and quality of life outcomes. Psychooncology. 2003 Jun;12(4):357-74. doi: 10.1002/pon.658. PMID 12748973
- [Result] Segal R, Evans W, Johnson D, Smith J, Colletta S, Gayton J, Woodard S, Wells G, Reid R. Structured exercise improves physical functioning in women with stages I and II breast cancer: results of a randomized controlled trial. J Clin Oncol. 2001 Feb 1;19(3):657-65. doi: 10.1200/JCO.2001.19.3.657. PMID 11157015
- [Result] Mock V, Frangakis C, Davidson NE, Ropka ME, Pickett M, Poniatowski B, Stewart KJ, Cameron L, Zawacki K, Podewils LJ, Cohen G, McCorkle R. Exercise manages fatigue during breast cancer treatment: a randomized controlled trial. Psychooncology. 2005 Jun;14(6):464-77. doi: 10.1002/pon.863. PMID 15484202
- [Result] Demark-Wahnefried W, Clipp EC, Morey MC, Pieper CF, Sloane R, Snyder DC, Cohen HJ. Lifestyle intervention development study to improve physical function in older adults with cancer: outcomes from Project LEAD. J Clin Oncol. 2006 Jul 20;24(21):3465-73. doi: 10.1200/JCO.2006.05.7224. PMID 16849763
- [Result] Coyne JC, Lepore SJ, Palmer SC. Efficacy of psychosocial interventions in cancer care: evidence is weaker than it first looks. Ann Behav Med. 2006 Oct;32(2):104-10. doi: 10.1207/s15324796abm3202_5. PMID 16972805
- [Result] Moadel AB, Shah C, Wylie-Rosett J, Harris MS, Patel SR, Hall CB, Sparano JA. Randomized controlled trial of yoga among a multiethnic sample of breast cancer patients: effects on quality of life. J Clin Oncol. 2007 Oct 1;25(28):4387-95. doi: 10.1200/JCO.2006.06.6027. Epub 2007 Sep 4. PMID 17785709
- [Result] Eversley R, Estrin D, Dibble S, Wardlaw L, Pedrosa M, Favila-Penney W. Post-treatment symptoms among ethnic minority breast cancer survivors. Oncol Nurs Forum. 2005 Mar 5;32(2):250-6. doi: 10.1188/05.ONF.250-256. PMID 15759063
- [Result] Northouse LL, Caffey M, Deichelbohrer L, Schmidt L, Guziatek-Trojniak L, West S, Kershaw T, Mood D. The quality of life of African American women with breast cancer. Res Nurs Health. 1999 Dec;22(6):449-60. doi: 10.1002/1098-240x(199912)22:63.0.co;2-a. PMID 10630287
- [Result] Ashing-Giwa KT, Padilla G, Tejero J, Kraemer J, Wright K, Coscarelli A, Clayton S, Williams I, Hills D. Understanding the breast cancer experience of women: a qualitative study of African American, Asian American, Latina and Caucasian cancer survivors. Psychooncology. 2004 Jun;13(6):408-28. doi: 10.1002/pon.750. PMID 15188447
- [Result] Watson M, Homewood J, Haviland J, Bliss JM. Influence of psychological response on breast cancer survival: 10-year follow-up of a population-based cohort. Eur J Cancer. 2005 Aug;41(12):1710-4. doi: 10.1016/j.ejca.2005.01.012. PMID 16098457
- [Result] Cramp F, Daniel J. Exercise for the management of cancer-related fatigue in adults. Cochrane Database Syst Rev. 2008 Apr 16;(2):CD006145. doi: 10.1002/14651858.CD006145.pub2. PMID 18425939
- [Result] Ballard-Barbash R, Friedenreich CM, Courneya KS, Siddiqi SM, McTiernan A, Alfano CM. Physical activity, biomarkers, and disease outcomes in cancer survivors: a systematic review. J Natl Cancer Inst. 2012 Jun 6;104(11):815-40. doi: 10.1093/jnci/djs207. Epub 2012 May 8. PMID 22570317
- [Result] Lof M, Bergstrom K, Weiderpass E. Physical activity and biomarkers in breast cancer survivors: a systematic review. Maturitas. 2012 Oct;73(2):134-42. doi: 10.1016/j.maturitas.2012.07.002. Epub 2012 Jul 26. PMID 22840658
- [Result] Long Parma D, Hughes DC, Ghosh S, Li R, Trevino-Whitaker RA, Ogden SM, Ramirez AG. Effects of six months of Yoga on inflammatory serum markers prognostic of recurrence risk in breast cancer survivors. Springerplus. 2015 Mar 26;4:143. doi: 10.1186/s40064-015-0912-z. eCollection 2015. PMID 25853030
- [Result] Mittra I, Khare NK, Raghuram GV, Chaubal R, Khambatti F, Gupta D, Gaikwad A, Prasannan P, Singh A, Iyer A, Singh A, Upadhyay P, Nair NK, Mishra PK, Dutt A. Circulating nucleic acids damage DNA of healthy cells by integrating into their genomes. J Biosci. 2015 Mar;40(1):91-111. doi: 10.1007/s12038-015-9508-6. PMID 25740145
- [Result] Mittra I, Samant U, Sharma S, Raghuram GV, Saha T, Tidke P, Pancholi N, Gupta D, Prasannan P, Gaikwad A, Gardi N, Chaubal R, Upadhyay P, Pal K, Rane B, Shaikh A, Salunkhe S, Dutt S, Mishra PK, Khare NK, Nair NK, Dutt A. Cell-free chromatin from dying cancer cells integrate into genomes of bystander healthy cells to induce DNA damage and inflammation. Cell Death Discov. 2017 May 29;3:17015. doi: 10.1038/cddiscovery.2017.15. eCollection 2017. PMID 28580170
- [Result] Andrykowski MA, Curran SL, Lightner R. Off-treatment fatigue in breast cancer survivors: a controlled comparison. J Behav Med. 1998 Feb;21(1):1-18. doi: 10.1023/a:1018700303959. PMID 9547419